CLINICAL TRIAL: NCT02961946
Title: Effects of Sublingual and Transdermal Administration of Nitroglycerin for Coronary CT Angiography on Image Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian Ghoshhajra, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016P002417
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sublingual Nitroglycerin spray (Active Comparator): Sublingual Nitroglycerin spray of 0.8 mg
  Interventions: Drug: Nitroglycerin
- Sublingual Nitroglycerin tablet (Active Comparator): Sublingual Nitroglycerin tablet of 0.8 mg
  Interventions: Drug: Nitroglycerin
- Nitroglycerin skin patch (Active Comparator): Nitroglycerin skin patch of 0.8 mg/h
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — Patients grouped in sublingual administration (group 1 and 2) will receive Nitroglycerin during the cCTA scan by the MD after the Calcium scoring scan and 5 minutes before the actual cCTA scan. Patients categorized to transdermal administration will receive Nitroglycerin 1 hour before the CT examination. The patch will be placed on the chest or the upper arm.

SUMMARY:
To evaluate image quality of coronary CT angiography (cCTA) after sublingual and transdermal administration of Nitroglycerin. Aim of this prospective research study is to investigate equivalence on image quality after sublingual or transdermal Nitroglycerin administration (H0).

Furthermore, the feasibility of transdermal Nitroglycerin administration will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled cCTA with contrast.
2. Able to comprehend and sign the consent form.

Exclusion Criteria:

1. Known hypersensitivity to glyceryl trinitrate, and related organic nitrates.
2. Acute circulatory failure associated with marked hypotension (shock).
3. Conditions associated with elevated intracranial pressure, cerebral haemorrhage and head trauma.
4. Closed-angle glaucoma.
5. Phosphodiesterase type 5 (PDE5) inhibitors such as sildenafil (Viagra®), tadalafil (Cialis), or vardenafil (Levitra) within the last 24 hours
6. Unstable clinical conditions (i.e. hemodynamic instability, arrhythmias)
7. Critical aortic stenosis
8. Systolic blood pressure < 90 mmHg
9. Pregnant or lactating female; premenopausal women with a positive urine pregnancy test.
10. Age under 18
11. Unwilling or unable to inform consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sublingual Nitroglycerin Spray | Sublingual Nitroglycerin Tablet | Nitroglycerin Skin Patch
Started | 66 | 66 | 66
Completed | 66 | 66 | 66
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Nitroglycerin Spray | Sublingual Nitroglycerin Tablet | Nitroglycerin Skin Patch | Total
Number analyzed (Participants) | 66 | 66 | 66 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 58 (13) | 57 (12) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 35 | 91
  Male | 34 | 42 | 31 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Coronary diameter [Mean (Standard Deviation); unit: mm] | 3.3 (0.9) | 3.5 (1.0) | 3.4 (1.0) | 3.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Coronary Artery Diameter Change
Description: Average diameter of coronary arteries at 7 predefined locations in the proximal, mid, and distal segments of the left main, left anterior descending, left circumflex and right coronary artery. Measurements avoid areas of coronary non-calcified and calcified plaques and measured twice for each location. Proximal and distal deviation from original measurements is possible in case of plaque.
Time Frame: obtained on the same day (day 0) of nitroglycerine administration (nitroglycerine is administered during the cCTA exam appointment).
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Sublingual Nitroglycerin Spray | Sublingual Nitroglycerin Tablet | Nitroglycerin Skin Patch
Number analyzed (Participants) | 66 | 66 | 66
Fold change | 1.14 [1.12 to 1.15] | 1.13 [1.09 to 1.16] | 1.15 [1.13 to 1.18]

ADVERSE EVENTS:
Time Frame: From time of nitroglycerin was given until until patients left the Radiology department. Usually 1 hour after the exam.
Description: There were no patients with serious adverse events. There were no patients with all-cause mortality. There were no patients with other adverse events.
Groups:
- Sublingual Nitroglycerin Spray: Sublingual Nitroglycerin spray of 0.8 mg
  Patients will receive Nitroglycerin during the cCTA scan by the MD after the Calcium scoring scan and 5 minutes before the actual cCTA scan.
- Sublingual Nitroglycerin Tablet: Sublingual Nitroglycerin tablet of 0.8 mg
  Patients will receive Nitroglycerin during the cCTA scan by the MD after the Calcium scoring scan and 5 minutes before the actual cCTA scan.
- Nitroglycerin Skin Patch: Nitroglycerin skin patch of 0.8 mg/h
  Patients categorized to transdermal administration will receive Nitroglycerin after Calcium scoring scan and 1 hour before the cCTA examination. The patch will be placed on the chest or the upper arm.
Arm/Group | Sublingual Nitroglycerin Spray | Sublingual Nitroglycerin Tablet | Nitroglycerin Skin Patch
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66 | 0/66

LIMITATIONS AND CAVEATS:
To evaluate coronary diameter change by nitroglycerin administration, non-constrast and contrast ECG-gated images were compared. Measurements avoided areas of visible arteriosclerosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT02961946/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT02961946/ICF_001.pdf